CLINICAL TRIAL: NCT06656052
Title: To Determine the Effects of Different Types of Cognitive Loading on Gait With Growing Age
Brief Title: Effects of Different Types of Cognitive Loading on Gait With Growing Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: REC/01884 Imran Amjad
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Gait Analysis; Cognitive Load, Performance
Keywords: gait; cognitive load; cognitive loading

STUDY DESIGN:
Intervention Model Description: research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First Age Group (Experimental): Participants with Age 21-30 years. All members of group number 1 who fall in the eligibility criteria will undergo three different types of cognitive loading. Three types of cognitive loading will be applied randomly to eliminate any bias. Each Method will be used three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. working memory task.; Other: 2. Visual and Verbal Fluency Task; Other: 3. Motor Task
- Second Age Group (Experimental): Participants with age 31-40 years. All members of group number 2 who fall in the eligibility criteria will undergo three different types of cognitive loading. Three types of cognitive loading will be applied randomly to eliminate any bias. Each Method will be used three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. working memory task.; Other: 2. Visual and Verbal Fluency Task; Other: 3. Motor Task
- Third Age Group (Experimental): Participants with Age 41-50 years. All members of group number 3 who fall in the eligibility criteria will undergo three different types of cognitive loading. Three types of cognitive loading will be applied randomly to eliminate any bias. Each Method will be used three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. working memory task.; Other: 2. Visual and Verbal Fluency Task; Other: 3. Motor Task
- Fourth Age Group (Experimental): Participants with age 51-60 years. All members of group number 4 who fall in the eligibility criteria will undergo three different types of cognitive loading. Three types of cognitive loading will be applied randomly to eliminate any bias. Each Method will be used three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. working memory task.; Other: 2. Visual and Verbal Fluency Task; Other: 3. Motor Task
- Fifth Age Group (Experimental): Participants with age 61-70 years. All members of group number 5 who fall in the eligibility criteria will undergo three different types of cognitive loading. Three types of cognitive loading will be applied randomly to eliminate any bias. Each Method will be used three times with pre and post-recordings to ensure reliability.
  Interventions: Other: 1. working memory task.; Other: 2. Visual and Verbal Fluency Task; Other: 3. Motor Task

INTERVENTIONS:
Other: 1. working memory task. — Arithmetic test (Backward counting with serial 3 subtraction and articulation): participants will be asked to count out loud backward with serial subtraction of 3 from each number, starting with a random number provided by the researcher.
Other: 2. Visual and Verbal Fluency Task — Stroop colour word test (modified Stroop test): participants will be asked to name the colour of ink that each word is printed in. This test will appear on the mobile phone in their hands while they walk to increase the effect of cognitive loading.
Other: 3. Motor Task — Participants will be asked to hold a tray of glasses filled with water and walk 10 meters to calculate the effect of cognitive loading on gait.

SUMMARY:
The goal of this study is to determine how different types of cognitive loading affect the gait of an individual and its association with growing age. The main aim is to find out if:

1. There is a significant difference in the effect of three different methods of cognitive loading on gait parameters across age groups.
2. There is an association of cognitive loading with different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female genders.
* Age between 21-70 years.
* Healthy individuals with normal systemic history.
* Individuals with normal cognitive level (score between 0-7 on 6CIT test)

Exclusion Criteria:

* Individuals having any comorbidities.
* Individuals having diagnosed gait disorders/deviations.
* Non-cooperative participants

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Walking speed | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the walking speed of the participant. A decrease in walking speed is the usual effect of cognitive loading on this gait parameter.
Walking speed | During three cognitive tasks
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the walking speed of the participant. A decrease in walking speed is the usual effect of cognitive loading on this gait parameter.
Walking speed | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the walking speed of the participant. A decrease in walking speed is the usual effect of cognitive loading on this gait parameter.
Gait Symmetry | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the gait symmetry of the participant. A decrease in gait symmetry is the usual effect of cognitive loading on this gait parameter.
Gait Symmetry | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the gait symmetry of the participant. A decrease in gait symmetry is the usual effect of cognitive loading on this gait parameter.
Gait Symmetry | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the gait symmetry of the participant. A decrease in gait symmetry is the usual effect of cognitive loading on this gait parameter.
Step length | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length of the participant. An increase in step length is the usual effect of cognitive loading on this gait parameter.
Step length | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length of the participant. An increase in step length is the usual effect of cognitive loading on this gait parameter.
Step length | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length of the participant. An increase in step length is the usual effect of cognitive loading on this gait parameter.
Step length variability | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length variability of the participant. An increase in step length variability is the usual effect of cognitive loading on this gait parameter.
Step length variability | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length variability of the participant. An increase in step length variability is the usual effect of cognitive loading on this gait parameter.
Step length variability | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length variability of the participant. An increase in step length variability is the usual effect of cognitive loading on this gait parameter.
Step time | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time of the participant. An increase in step time is the usual effect of cognitive loading on this gait parameter.
Step time | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time of the participant. An increase in step time is the usual effect of cognitive loading on this gait parameter.
Step time | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time of the participant. An increase in step time is the usual effect of cognitive loading on this gait parameter.
Step time variability | Baseline
  Smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time variability of the participant. An increase in step time variability is the usual effect of cognitive loading on this gait parameter.
Step time variability | During Cognitive loading tests
  Smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time variability of the participant. An increase in step time variability is the usual effect of cognitive loading on this gait parameter.
Step time variability | Immediately after Cognitive loading tests
  Smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time variability of the participant. An increase in step time variability is the usual effect of cognitive loading on this gait parameter.
Step length asymmetry | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length asymmetry of the participant. An increase in step length asymmetry is the usual effect of cognitive loading on this gait parameter.
Step length asymmetry | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length asymmetry of the participant. An increase in step length asymmetry is the usual effect of cognitive loading on this gait parameter.
Step length asymmetry | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step length asymmetry of the participant. An increase in step length asymmetry is the usual effect of cognitive loading on this gait parameter.
Step time asymmetry | Baseline
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time asymmetry of the participant. An increase in step time asymmetry is the usual effect of cognitive loading on this gait parameter.
Step time asymmetry | During Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time asymmetry of the participant. An increase in step time asymmetry is the usual effect of cognitive loading on this gait parameter.
Step time asymmetry | Immediately after Cognitive loading tests
  A smartphone-based accelerometer through a mobile app named Gait & Balance (G&B app) will be used to detect the step time asymmetry of the participant. An increase in step time asymmetry is the usual effect of cognitive loading on this gait parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No